CLINICAL TRIAL: NCT05583747
Title: Electrical Field Modeling to Engage Neurophysiological Targets of Intermittent Theta Burst Stimulation in Treatment Resistant Depression (E-Fields iTBS)
Brief Title: E-field Guided iTBS for Treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3773
Record Dates: First submitted 2022-06-08; First posted 2022-10-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder
Keywords: brain stimulation; rTMS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Course A: E-field Modeling (Experimental): Your Magnetic Resonance Image (MRI) results and rTMS calibration information (motor threshold) will be used to create a brain model and identify the targeted location, iTBS coil position and intensity for your iTBS rTMS treatment. You will undergo iTBS rTMS treatment in this study for 6 weeks. There will be 5 iTBS treatment sessions per week, lasting approximately 3 minutes each, once daily for 5 days in a row (always Monday to Friday). Each day after treatment, you will also complete a brief set of questionnaires to track your symptoms, which will take 15 minutes. After every 5 treatments, you will complete an extra interview that will take an additional 30 minutes. There will also be two follow-up visits at 1 and 4 weeks after the end of treatment, each lasting approximately 1 hour. During these follow-up visits, you will be asked to complete a brief set of questionnaires and interviews to monitor your symptoms.
  Interventions: Device: iTBS
- Treatment Course B: Beam F3 (Active Comparator): The targeted iTBS rTMS treatment location and intensity will be determined via standard parameters, specifically anatomical landmarks and your rTMS calibration information (motor threshold). You will undergo iTBS rTMS treatment in this study for 6 weeks. There will be 5 iTBS treatment sessions per week, lasting approximately 3 minutes each, once daily for 5 days in a row (always Monday to Friday). Each day after treatment, you will also complete a brief set of questionnaires to track your symptoms, which will take 15 minutes. After every 5 treatments, you will complete an extra interview that will take an additional 30 minutes. There will also be two follow-up visits at 1 and 4 weeks after the end of treatment, each lasting approximately 1 hour. During these follow-up visits, you will be asked to complete a brief set of questionnaires and interviews to monitor your symptoms.
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — rTMS involves direct stimulation of cortical neurons using externally applied, powerful, focused magnetic field pulses. iTBS is a briefer form of patterned rTMS that has been shown to be effective against MDD, despite a stimulation period of 1-3 min rather than 30-40 min.

SUMMARY:
The purpose of this study is to establish how personalization of repetitive transcranial magnetic stimulation (rTMS) can change markers of brain activity and improve treatment response. To do this, all participants will receive the same active form of treatments, but some of the participants in this study will receive intermittent theta burst stimulation (iTBS) rTMS treatment with standard forms of targeting and intensity, and others will receive iTBS rTMS treatment using personalized magnetic resonance imaging (MRI) and electric field (E-field) modeling measures.

DETAILED DESCRIPTION:
The purpose of this study is to establish how personalization of rTMS can change markers of brain activity and improve treatment response in major depressive disorder (MDD). All participants will receive up to 30 iTBS treatments to the left dorsolateral prefrontal cortex (DLPFC), delivered daily, 5 days per week, for 6 weeks. Participants will be randomized to either a standard treatment arm, in which the iTBS targeting will be via the Beam F3 method to identify the left DLPFC location, and intensity will be determined as 120% of the resting motor threshold, or a personalized arm, in which the left DLPFC will be identified via functional magnetic resonance imaging (fMRI), the optimal coil position and stimulus intensity will be derived through E-Field modeling pipelines.

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients;
2. are voluntary and competent to consent to treatment;
3. have a Diagnostic and Statistical Manual for Mental Disorders, 5th edition major depressive episode based on the Mini International Neuropsychiatric Interview (MINI)
4. are 18yo to 65yo;
5. have a score of ≥18 on the Hamilton Rating Scale for Depression (HRSD-17) item at screening
6. have not had a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of ≥ 3 in the current episode or have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2);
7. are agreeable to keeping their current medication constant during the study
8. are able to adhere to the study and treatment schedules
9. meet TMS and MRI safety criteria

Exclusion Criteria:

1. have a concomitant unstable medical illness
2. are pregnant or intend to become pregnant during the study
3. have a current MINI diagnosis of bipolar disorder, psychotic disorder, obsessive compulsive disorder, concurrent substance use disorder (aside from nicotine) or post-traumatic stress disorder (current or within the last year)
4. have failed a course of electroconvulsive therapy within the current depressive episode due to the lower likelihood of response to rTMS;
5. have any significant neurological disorder (e.g., space occupying brain lesion, history of stroke, cerebral aneurysm, seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis) or confirmed diagnosis of dementia or cognitive impairment
6. present with a medical condition, medication, or laboratory abnormality that could cause a major depressive episode in the opinion of the investigator
7. have an intracranial implant or any other metal object that cannot be safely removed, precluding safety of TMS or MRI exposure within or near the head, excluding the mouth
8. require benzodiazepine equivalent to lorazepam 2 mg/day or higher or any anticonvulsant due to the potential of these medications to limit the efficacy of rTMS [45]
9. have inadequate English fluency to complete clinical assessments.
10. are participating in a new course psychotherapy initiated within the last 3 months or finishing prior to the end of scheduled treatments;
11. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Markers of cortical excitation | change from pre-intervention to post-intervention (average of 6 weeks)
  TMS-EEG markers of increased cortical excitation (GMFA-AUC)
Depression scores | changes from baseline to Week 4 follow-up
  Hamilton depression rating scale (HDRS-17) scores

SECONDARY OUTCOMES:
Peripheral biomarkers | change from Pre- and post-intervention (average of 6 weeks)
  Circulating volumes of gamma-aminobutyric acid (GABA), brain-derived neurotrophic factor (BDNF) and N-methyl-D-aspartate (NMDA) proteins

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Poul Hansen Family Centre for Depression, Toronto Western Hospital, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario